CLINICAL TRIAL: NCT07162714
Title: Short-Course Radiotherapy Followed by Ivonescimab (AK112) in pMMR/MSS Mid-Low Rectal Cancer: An Exploratory Phase II Clinical Study.
Brief Title: SCRT Followed by AK112 in pMMR/MSS Mid-low Rectal Cancer
Acronym: STAR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Akeso (Industry)
Responsible Party: Principal Investigator, Ji Zhu, Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR
Record Dates: First submitted 2025-03-07; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer; Radiation; AK112
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): The patients receive pelvic radiotherapy: Intensity-Modulated Radiation Therapy (IMRT) or Volumetric Modulated Arc Therapy (VMAT), with a total dose of 25 Gy delivered in 5 fractions. One week post-radiotherapy, treatment with Ivonescimab (AK112) was initiated at a dose of 20 mg/kg via intravenous infusion on Day 1 of each 21-day cycle, for a total of 6 cycles.
  Treatment response was assessed after 3 cycles. Patients with Progressive Disease (PD) were withdrawn from the study and promptly switched to alternative regimens.
  Patients achieving CR/PR/SD continued treatment for an additional 3 cycles.A comprehensive evaluation was conducted after completing 6 cycles. Patients achieving clinical Complete Response (cCR) were eligible for watchful waiting. For those not attaining cCR, Total Mesorectal Excision (TME) surgery was recommended. The need for adjuvant chemotherapy was subsequently determined based on postoperative pathological findings.
  Interventions: Radiation: radiotherapy; Drug: Ivonescimab (20mg/kg Q3W); Other: Non-operative Management; Procedure: Surgery

INTERVENTIONS:
Radiation: radiotherapy — The patients receive pelvic radiotherapy: Intensity-Modulated Radiation Therapy (IMRT) or Volumetric Modulated Arc Therapy (VMAT), with a total dose of 25 Gy delivered in 5 fractions. Radiotherapy is to start on day 1 and to finish on day 5.
Drug: Ivonescimab (20mg/kg Q3W) — The first dose of vonescimab (AK112) was administered 1 week after the completion of radiotherapy. Ivonescimab (AK112) was initiated at a dose of 20 mg/kg via intravenous infusion on Day 1 of each 21-day cycle, for a total of 6 cycles.
Other: Non-operative Management — Subjects who achieve cCR after radiation and 6 cycles treatment of Ivonescimab can, after discussion with the local investigator, decline surgery and opt for a non-operative management.
Procedure: Surgery — For patients who do not achieve cCR at the end of 6 cycles treatment of Ivonescimab, TME surgery is recommended.

SUMMARY:
Primary Objectives： Evaluate the complete response rate (CR rate) and safety of short - course radiotherapy combined with ivonesimab (AK112) in patients with pMMR/MSS mid - low rectal cancer.

Secondary Objectives： Evaluate treatment - related toxic reactions, the quality of life, long - term prognosis (local control [LC], disease - free survival [DFS] and overall survival [OS]).

Patients will :

Receive Radiotherapy: Pelvic IMRT or VMAT, DT 25Gy/5Fx. One week after radiotherapy, begin treatment with Ivorsimab (AK112) at a dose of 20mg/kg by intravenous drip on day 1. One cycle is 21 days, and a total of 6 cycles are to be carried out.

Evaluate the curative effect after 3 cycles of treatment. Patients with progressive disease (PD) will withdraw from the study, and other treatment plans will be adjusted in a timely manner. Patients with CR/PR/SD will continue treatment for another 3 cycles. Conduct a comprehensive assessment after 6 cycles of treatment. Patients who achieve cCR can choose the watch - and - wait approach. For patients who do not achieve cCR, TME surgery is recommended. Decide whether to perform adjuvant chemotherapy based on the postoperative pathological findings.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old;
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 - 1;
3. Histopathologically confirmed rectal adenocarcinoma, without any prior anti - tumor treatment; The status of MMR/MSI is detected by IHC/PCR in pathological biopsy to clarify that the patient's classification is pMMR/MSS;
4. The lower border of the lesion is ≤ 7 cm from the anal verge as determined by fibrocolonoscopy or digital rectal examination;
5. Baseline magnetic resonance staging is cT2 - 4 and/or N+, excluding any of cT4b, N2, positive mesorectal fascia (MRF+), extramural venous invasion (EMVI+), lateral lymph node metastasis, and distant metastasis (according to the 8th edition of the AJCC Cancer Staging Manual);
6. Able to accept the treatment plan during the study period;
7. Signed written informed consent.

Exclusion Criteria:

1. Uncontrolled epilepsy, history of central nervous system disorders or psychiatric conditions that, in the investigator's judgment, may interfere with the ability to provide informed consent or affect compliance with oral medication.
2. Prior immunotherapy for any indication or a history of severe hypersensitivity reactions to other monoclonal antibodies.
3. Clinically significant active cardiac disease, including symptomatic coronary artery disease, congestive heart failure (New York Heart Association [NYHA] Class II or higher), severe arrhythmias requiring medication, or a history of myocardial infarction within the past 12 months.
4. Immunosuppressive therapy following organ transplantation.
5. History of other malignancies within the past 5 years (excluding adequately treated non-melanoma skin cancer or carcinoma in situ).
6. Severe uncontrolled recurrent infections or other significant uncontrolled comorbidities.
7. Baseline laboratory values failing to meet the following criteria:Hemoglobin ≥80 g/L; Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelets ≥100×10^9/L; ALT/AST ≤2.5×upper limit of normal (ULN); Alkaline phosphatase (ALP) ≤2.5×ULN; Total bilirubin <1.5×ULN; Serum creatinine <1×ULN
8. Active gastrointestinal diseases (e.g., gastric/duodenal ulcers, ulcerative colitis), unresected tumors with active bleeding, or other conditions deemed by the investigator to pose risks of gastrointestinal bleeding or perforation.
9. Active bleeding or bleeding predisposition.
10. Pregnancy or lactation.
11. Hypersensitivity to any component of the investigational drug(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR rate) | at the end of 6 cycles of AK112 treatment (each cycle is 21 days) or after surgery
  including clinical complete response rate (cCR) and pathological complete response rate (pCR). pCR status is defined as the absence of resected speci mens with surviving tumour cells. cCR is defined as undetectable signs of tumour at least 4 weeks after TNT completion by clinical ex amination, including magnetic resonance imaging (MRI), endoscopy, digital rectal examination (DRE) and Positron Emission Tomography-Computed Tomography (PET-CT).

SECONDARY OUTCOMES:
Treatment - related adverse reactions | From enrollment to 6 months after the last administration of study treatment
  Number of Participants with Treatment - related adverse reactions according to CTCAE 5.0
locoregional control rate | Up to 3 years after the last administration of study treatment
  from the date of registration to the date of occurrence of locoregional recurrence, or death due to any cause.
disease-free survival rate | Up to 3 years after the last administration of study treatment
  from the date of registration to the date of occurrence of any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause.
Overall survival rate | Up to 3 years after the last administration of study treatment
  from the date of registration to the date of death from any cause.
Qol EORTC-C30 questionnaire | From enrollment to 6 months after the last administration of study treatment
Qol EORTCQLQ- CR29 questionnaire | From enrollment to 6 months after the last administration of study treatment